CLINICAL TRIAL: NCT03313544
Title: Evolution of the Heart Function When Monitoring Immunotherapies Anti-cancerous Inhibiting Programmed Cell Death 1 (PD-1)
Brief Title: Evolution of the Heart Function When Monitoring Immunotherapies Anti-cancerous Inhibiting PD-1
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-01; 2017-001197-42 (EudraCT Number)
Record Dates: First submitted 2017-10-10; First posted 2017-10-18 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Melanoma; Non-small Cell; Lung Cancer
MeSH Terms: conditions — Melanoma; Lung Neoplasms | interventions — Nivolumab; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NIVOLUMAB PATIENTS (Experimental)
  Interventions: Drug: Nivolumab; Device: MRI; Biological: BLOOD SAMPLES; Device: trans-thoracic echocardiography

INTERVENTIONS:
Drug: Nivolumab — NIVOLUMAB
Device: MRI — Cardiac MRI 6 MONTHS
Biological: BLOOD SAMPLES — biological (BNP and troponin)
Device: trans-thoracic echocardiography — 1, 3 and 6 months

SUMMARY:
Prospective, monocentric clinical study. Patients selected for nivolumab therapy in AP-HM for melanoma and non-small cell lung cancer will be eligible. Do not include patients with conditions that do not allow MRI, prior cardiovascular disease with LVEF<50%, cardiomyopathy, history of cardiac arrhythmia, history of cardiovascular toxicity under anticancer therapy, coronary artery disease or stroke less than 3 months Therapeutic management will not be modified and treatment will be administrated as usual.

Cardiovascular follow up will be identical to that recommended and realized in current care in the Cardio-Oncology unit of AP-HM. It will include clinical, biological (BNP and troponin) and trans-thoracic echocardiography (TTE) at baseline and then at 1, 3 and 6 months. Auto-antibodies against troponin I assay will be performed to avoid false negatives of normal blood level of troponin I at baseline and then at 6 months. Cardiac MRI will be performed as well at baseline and at the end of the study (6 months). MRI is the gold standard for ventricular function evaluation.

Primary endpoint will be left ventricular function evolution evaluated by global longitudinal strain (GLS, 2D speckles tracking) in TTE. Secondary endpoints will be left and right ventricular function parameters: LEVF by TTE and MRI, left ventricular indexed volumes by TTE and MRI, right ejection ventricular function and indexed volumes by TTE and MRI, systolic pulmonary arterial pressure by TTE, serum troponin I and BNP, arrhythmias and conduction disorders on the electrocardiogram (ECG).

Number of required subjects: GLS is recommended for following up left ventricular function under anticancer treatments. Based on the hypothesis of a significant GLS decrease (15%) in 20% of cases with alpha risk of 0.05 and accuracy of 0.12 which means expected confidence interval of 0.08-0.32, then the number of required subjects is 50 patients.

The inclusion period will be 18 months with a follow up if 6 months, ie a total duration of the study of 24 months.

ELIGIBILITY:
Inclusion Criteria:

patients treated with nivolumab

Exclusion Criteria:

* Age <18 years
* Preliminary cardiac disease with FeVG <50%
* Cardiomyopathy dilated, hypertrophic or restrictive
* History of cardiac arrhythmia
* History of cardiac toxicity under another anti-cancer treatment
* Known coronary disease
* History of stroke less than 3 months old
* Patient not wishing to participate in the study
* Vulnerable persons (pregnant women, adults under guardianship or guardianship, persons deprived of their liberty)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-04-09 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
systolic pulmonary arterial pressure | 6 months
  trans-thoracic echocardiography

SECONDARY OUTCOMES:
ventricular function evaluation. | 6 MONTHS
  MRI
serum troponin I | 1,3, 6 months
  BLOOD SAMPLES
Brain natriuretic peptide (BNP) | 1,3, 6 months
  BLOOD SAMPLES

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Study Director — assistance publique hôpitaux de marseille
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France

REFERENCES:
- [Derived] Cadour F, Cautela J, Rapacchi S, Varoquaux A, Habert P, Arnaud F, Jacquier A, Meilhac A, Paganelli F, Lalevee N, Scemama U, Thuny F. Cardiac MRI Features and Prognostic Value in Immune Checkpoint Inhibitor-induced Myocarditis. Radiology. 2022 Jun;303(3):512-521. doi: 10.1148/radiol.211765. Epub 2022 Mar 1. PMID 35230185